CLINICAL TRIAL: NCT01813058
Title: The Efficacy of Intravenous Tranexamic Acid in Decreasing Blood Loss in Pediatric Idiopathic Scoliosis Surgery?
Brief Title: Does Tranexamic Acid Decrease Blood Loss in Pediatric Idiopathic Scoliosis Surgery?
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Susan Goobie, Assistant in Anesthesia, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRB-P00003400
Record Dates: First submitted 2013-02-25; First posted 2013-03-18 (Estimated); Results first posted 2019-02-20 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2019-01

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: Tranexamic acid, Blood loss
MeSH Terms: conditions — Hemorrhage | interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo ( 0.9% Normal saline) intravenously given as a 0.5 ml/kg loading dose over 15 minutes followed by a 0.1 ml/kg/hr continuous infusion throughout the surgery.
  Interventions: Drug: Placebo
- Tranexamic acid (Active Comparator): Tranexamic acid 100 mg/ml; 50 mg/kg loading dose = 0.5 ml/kg LD given over 15 minutes and 10 mg/kg/hr = 0.1 ml/kg/hr infusion for the duration of the surgery.
  Interventions: Drug: Tranexamic Acid

INTERVENTIONS:
Drug: Tranexamic Acid — Following a standardized general anesthetic protocol, patients coming with idiopathic scoliosis will be randomized to either:
  1. placebo i.e. saline 0.9% (intravenous injection)
  2. intravenous TXA given as a loading dose over 15 minutes of 50 mg/kg bolus ( within an hour prior to surgical incision) and 10 mg/kg/hr infusion for the duration of the surgery.
  Other Names: Cyklokapron, TXA, TA
  Arms: Tranexamic acid
Drug: Placebo — Following a standardized general anesthetic protocol, patients coming with idiopathic scoliosis will be randomized to:
  1. Placebo ( 0.9% Normal saline) intravenously given as a 0.5 ml/kg loading dose over 15 minutes followed by a 0.1 ml/kg/hr continuous infusion throughout the surgery or
  2. TXA as previously described.
  Other Names: 0.9% Normal saline
  Arms: Placebo

SUMMARY:
Adolescent idiopathic scoliosis surgery is an extensive procedure associated with significant blood loss frequently requiring the transfusion of blood. Tranexamic acid (TXA) is a synthetic antifibrinolytic (prevents breakdown of the blood clot) that has been used to extensively reduce transfusion in pediatric major surgery, including cardiac, craniofacial and orthopedic surgery. In this prospective randomized double-blinded study, the investigators wish to evaluate the hypothesis that TXA is more effective than standard of care at decreasing blood loss and blood transfusion perioperatively in children and adolescents undergoing idiopathic scoliosis surgery.

DETAILED DESCRIPTION:
This prospective randomized double-blinded study will enroll 120 children and adolescents ages undergoing scoliosis repair with the diagnosis of idiopathic scoliosis. The primary aim is to determine if intravenous infusion of TXA is more effective than standard care (no TXA) at decreasing blood loss and blood transfusion perioperatively in children and adolescents presenting for scoliosis surgery.

Aims:

1. Investigate and compare the efficacy of TXA (as measured by intraoperative blood loss and blood transfusion) intravenously administered during surgery vs placebo in patients with idiopathic scoliosis coming for surgery.
2. Determine the PK profile of TXA in children and adolescents undergoing scoliosis surgery.
3. Investigate the contribution of these different factors (plasma concentration of TXA, age related differences in PK/PD and renal function, and polymorphism of the Plasminogen activator inhibitor-1 (PAI-1) gene and PAI-1 levels with TXA efficacy in pediatric patients undergoing and scoliosis surgery.
4. Determine the safety profile of intravenous TXA in children and adolescents presenting for scoliosis surgery.

Following a standardized general anesthetic protocol, patients coming with idiopathic scoliosis will be randomized to either:

1. placebo i.e. saline 0.9% (intravenous injection)
2. intravenous TXA given as a loading dose over 15 minutes of 50 mg/kg bolus ( 30- 60 minutes prior to surgical incision) and 10 mg/kg/hr infusion for the duration of the surgery.

During the surgery, we will follow standardized, defined fluid, blood and blood production management protocols.

The following data are part of routine patient care and will be collected for study purposes:

1. Age, weight, height, gender, race, coexisting diseases, preoperative hemoglobin, hematocrit, platelets, PT, PTT, and INR, creatinine.
2. Intraoperative data: total volume of intraoperative blood loss as estimated by weighing sponges amount of blood in suction canisters, total volumes and units of blood products administered, total volume of cell saver blood administered, total volumes of crystalloid and colloid agents administered, hemodynamic parameters; mean arterial blood pressure & heart rate, total urine output, total surgical time, and number spinal levels involved.
3. Laboratory data: Perioperative baseline and serial hemoglobin, hematocrit, platelet count, PT, PTT, INR and fibrinogen as dictated by standard clinical practice.
4. Postoperative data collection will include: blood transfusion requirement in the first 24 hours after surgery, amount of blood collected in the surgical drains for the first 24 hours postoperatively, the occurrence of any postoperative complications and duration of ICU and hospital stay.

A research team member will follow the patient daily after the surgery and a follow-up phone call will be made to the family at one month after discharge from the hospital with the aim to identify adverse events related to TXA. Potential adverse advents include hypersensitivity or allergic reaction to tranexamic acid, thromboembolic events, neurological complications, and development of renal insufficiency. Adverse events will be reported immediately to the IRB as per institutional protocols. As the estimate of blood loss is somewhat inaccurate, blood loss will also be calculated as previously described.

The following measures are not part of routine patient care but are required by the study protocol:

During the course of the operation, a total of four samples consisting of 2 ml each of blood will be drawn from the arterial catheter for DNA, PAI-1 protein level, and baseline TXA. After the study drug infusion is started, subsequent 2 ml samples will be drawn utilizing one of four different sampling schemes randomly assigned.

TXA plasma concentrations will be measured as described with some modifications we have made in our laboratory18. The samples will be immediately anticoagulated with ethylene diamine tetraacetic acid (EDTA) and stored on ice. Plasma will be separated by centrifugation (1000g x10 min at 4oC) and stored at -70 oC pending analysis for TXA concentrations. TXA plasma concentrations will be measured using high performance liquid chromatography (HPLC) after ultrafiltration and derivatization18.

Recruitment Methods:

Potential eligibility for the study will be identified via the surgical schedule which will be screened daily by a designated member of the research team. A cover letter, brochure, and consent form will be mailed to the prospective patient's family prior to the scheduled pre-operative appointment. The study protocol will be reviewed with the patient/family and all queries will be addressed on the day of the visit to the preoperative clinic prior to the scheduled date of surgery. Informed consent will be obtained from the parents/legal guardians as per institutional IRB guidelines. The child's assent (when appropriate) will also be obtained at least 24 hours before the scheduled surgery when possible.

Data Analysis Plan:

A preliminary power analysis indicated that a total sample size of 120 children randomized equally to TXA vs. standard of care (no TXA) will provide 80% power (α = 0.05, β = 0.20) to detect a decrease from 30% to 10% of patients loosing a significant amount of blood (defined as >/= 25 ml/kg) using a chi-square test of independent binomial proportions assuming a standard deviation of 25% (effect size = 1.2) (version 7.0, nQuery Advisor, Statistical Solutions, Saugus, MA).

Adverse Event Criteria and Reporting Procedures:

Potential adverse events include hypersensitivity or allergic reaction to tranexamic acid or any component, thromboembolic events, neurologic events such as seizures, hypotension (with rapid IV administration). In awake patients, the following has been reported: nausea, diarrhea or vomiting. The patients will be assessed the next day by a member of the research team and interviewed for the occurrence of any of these adverse events. In the event of a serious adverse event, it will be reported to the IRB immediately and the study halted until a thorough investigation into the cause can be made.

Data and Safety Monitoring Plan Data collection for this study will include the collection of any data pertaining to adverse events. Any adverse events will be promptly reported to the IRB and the members of the research team responsible for data and safety monitoring. Data and safety monitoring will be reviewed by the research team every 10 subjects recruited or earlier if a specific problem is identified

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents (age 10-21 yr) for elective Idiopathic scoliosis corrective surgery; posterior repair.

Exclusion Criteria:

* Preexisting coagulopathy, (INR>1.4, PTT>1.4xN, PT>1.4xN, platelet count<150,000/mm3), severe hematological disorders, hepatic failure, or renal failure. Ingestion of acetylsalicylate within 14 days or NSAIDs within 2 days of the scheduled surgery date; history of prior blood transfusion. Pre-donation of autologous blood. Patients having anterior-posterior repair.

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2013-01; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Goobie, MD, FRCPC, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Childrens Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sethna NF, Zurakowski D, Brustowicz RM, Bacsik J, Sullivan LJ, Shapiro F. Tranexamic acid reduces intraoperative blood loss in pediatric patients undergoing scoliosis surgery. Anesthesiology. 2005 Apr;102(4):727-32. doi: 10.1097/00000542-200504000-00006. PMID 15791100
- [Result] Goobie SM, Meier PM, Pereira LM, McGowan FX, Prescilla RP, Scharp LA, Rogers GF, Proctor MR, Meara JG, Soriano SG, Zurakowski D, Sethna NF. Efficacy of tranexamic acid in pediatric craniosynostosis surgery: a double-blind, placebo-controlled trial. Anesthesiology. 2011 Apr;114(4):862-71. doi: 10.1097/ALN.0b013e318210fd8f. PMID 21364458
- [Result] Goobie SM, Meier PM, Sethna NF, Soriano SG, Zurakowski D, Samant S, Pereira LM. Population pharmacokinetics of tranexamic acid in paediatric patients undergoing craniosynostosis surgery. Clin Pharmacokinet. 2013 Apr;52(4):267-76. doi: 10.1007/s40262-013-0033-1. PMID 23371895

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo ( 0.9% Normal saline) intravenously given as a 0.5 ml/kg loading dose over 15 minutes followed by a 0.1 ml/kg/hr continuous infusion throughout the surgery.
  Placebo: Following a standardized general anesthetic protocol, patients coming with idiopathic scoliosis will be randomized to:
  1. Placebo ( 0.9% Normal saline) intravenously given as a 0.5 ml/kg loading dose over 15 minutes followed by a 0.1 ml/kg/hr continuous infusion throughout the surgery or
  2. TXA as previously described.
- Tranexamic Acid: Tranexamic acid 100 mg/ml; 50 mg/kg loading dose = 0.5 ml/kg LD given over 15 minutes and 10 mg/kg/hr = 0.1 ml/kg/hr infusion for the duration of the surgery.
  Tranexamic Acid: Following a standardized general anesthetic protocol, patients coming with idiopathic scoliosis will be randomized to either:
  1. placebo i.e. saline 0.9% (intravenous injection)
  2. intravenous TXA given as a loading dose over 15 minutes of 50 mg/kg bolus ( within an hour prior to surgical incision) and 10 mg/kg/hr infusion for the duration of the surgery.
Period: Overall Study
Arm/Group | Placebo | Tranexamic Acid
Started | 60 | 60
Completed | 55 | 56
Not Completed | 5 | 4
Not completed — Withdrawal by Subject | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Tranexamic Acid | Total
Number analyzed (Participants) | 55 | 56 | 111
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 55 | 56 | 111
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.7 (1.8) | 14.9 (2.0) | 14.8 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 46 | 88
  Male | 13 | 10 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 43 | 46 | 89
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 9 | 5 | 14
weight [Mean (Standard Deviation); unit: kg] | 56.6 (11.9) | 55.1 (11.8) | 56 (11.8)
American Society of Anesthesiology Physical Status Classification [Median (Inter-Quartile Range); unit: units on a scale] — The ASA PHYSICAL STATUS CLASSIFICATION SYSTEM scale is 1-6, ASA 1 being the lowest risk and ASA4 being the higher risk as follows ( ASA 5 AND 6 DO NOT APPLY TO THIS POPULATION):
  ASA I A normal healthy patient ASA II A patient with mild systemic disease ASA III A patient with severe systemic disease ASA IV A patient with severe systemic disease that is a constant threat to life ASA V A moribund patient who is not expected to survive without the operation ASA VI A declared brain-dead patient whose organs are being removed for donor purposes
  units on a scale | 2 [1 to 3] | 2 [1 to 3] | 2 [1 to 3]

OUTCOME MEASURES:

1. Primary Outcome: Perioperative Blood Loss
Description: Perioperative blood loss (during operation and for entire hospital admission)
Time Frame: perioperarively - during entire hospital admission
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Placebo | Tranexamic Acid
Number analyzed (Participants) | 55 | 56
mL | 1031 (484) | 836 (373)
Statistical Analysis 1: Comparison: Placebo vs Tranexamic Acid; Test type: Superiority; p < 0.001, Fisher Exact; Mean Difference (Final Values) = 195

ADVERSE EVENTS:
Time Frame: during entire hospital admission up to seven days
Arm/Group | Placebo | Tranexamic Acid
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/56
Other Adverse Events (participants affected / at risk) | 0/55 | 0/56

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No